CLINICAL TRIAL: NCT03299205
Title: Alcohol & Metabolic Comorbidities in PLWHA: Evidence Driven Interventions
Acronym: ALIVE-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Patricia Molina, Professor and Head Department of Physiology, Louisiana State University Health Sciences Center in New Orleans
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9767
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: HIV/AIDS; Dysglycemia; Alcohol Use Disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcoholism | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Aerobic exercise program using treadmill.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention consists of moderate intensity aerobic exercise intervention that will include the wearing of an accelerometer (i.e. Fitbit Zip) to monitor daily activity and steps. Aerobic exercise will be conducted over 10-weeks in PLWHA +/- AUD. The programs will consist of aerobic exercise 3 days per week of moderate intensity for 30-45 minutes each session with the goal of achieving 135 minutes per week. The program will begin at low-moderate intensity and progress to higher intensity exercise after week 4 of the program. All exercise will be completed on a treadmill and supervised by study staff. Each participant will be provided with a Fitbit Zip to monitor daily activity and steps with a goal of 7000 steps per day.

SUMMARY:
Cross-sectional and prospective studies are proposed to test the prediction that a higher proportion of HIV+ individuals with hazardous alcohol drinking with subclinical fasting dysglycemia will present with impaired oral glucose tolerance and dysfunctional metabolic skeletal muscle phenotype. Prospective studies will test the efficacy of an exercise intervention in improving glycemic control. Results will inform larger scale interventions to ameliorate metabolic comorbidities, improve health, quality of life, and possibly decrease hazardous alcohol drinking.

DETAILED DESCRIPTION:
Adult male and female in care PLWHA with fasting plasma glucose (FPG) >94 mg/dL and <125 mg/dL will be recruited. Measures of FPG and HbA1c obtained from overnight fasted subjects. Alcohol use disorder (AUD) will be assessed by AUDIT and time-line follow back questionnaires, coupled with Phosphatidylethanol (PEth) measures. Glucose tolerance will be assessed by oral glucose tolerance test (OGTT). Blood sample collected at the time of the OGTT will be used for determination of circulating levels of adipokines (adiponectin and resistin).

A subset of adult male and female PLWHA +/- AUD with impaired OGTT will be recruited to undergo skeletal muscle (SKM) biopsy (vastus lateralis), 90 min after a defined (calorie and nutrient composition) meal (i.e.,Ensure, Carnation Instant Breakfast). Muscle samples will be used for phenotype characterization (markers of inflammation, insulin signaling, mitochondrial homeostasis) and for myoblast isolation.

Adult male and female PLWHA +/- AUD with impaired OGTT will undergo a moderate intensity aerobic exercise intervention that will include the wearing of an accelerometer (i.e. Fitbit Zip) to monitor daily activity and steps. A SKM biopsy will be performed after completion of the exercise protocol in a subset of subjects to examine the changes in gene expression and myoblast mitochondrial oxidative capacity. We will expand recruitment by enrolling PLWHA +/- AUD based on a FPG between 94-120 mg/dL to participate in the exercise intervention. Clearance for participation in this study will require EKG, completion of a physical activity readiness questionnaire, and medical clearance from a staff clinician. Individuals with significant peripheral neuropathies or the prevalence of significant cardiovascular impairments (i.e. resting cardiac abnormalities or arrhythmias, severe hypertension, etc.) will be excluded from exercise testing or intervention. The 10-week exercise intervention program will consist of aerobic exercise 3 days per week of moderate intensity for 30-45 minutes each session with the goal of achieving 135 minutes per week. The program will begin at low-moderate intensity (40 to 50% of heart rate reserve; HRR) and progress to a higher intensity (50 to 60% HRR) exercise after week 4 of the program. The frequency and duration of exercise sessions will remain constant after week 4 so the absolute dose of exercise will be altered through increasing intensity, i.e. from low-moderate to more vigorous. All exercise will be completed on a treadmill at the Louisiana State University Health Sciences Center (LSUHSC) Wellness Center. Additionally, each participant will be provided with a Fitbit Zip to monitor daily activity and steps. Data from the Fitbit Zip will be downloaded weekly basis. Participants will be given a healthy step goal of 7000 steps per day. Based on initial step counts after the first week of wearing the accelerometer, individual goals will be discussed with the participants. Personal limitations that develop during the study period (i.e. peripheral neuropathy, orthopedic limitation, etc.) will be monitored and will be reason for exclusion from the exercise program. All sessions will be supervised and adherence to the exercise prescription will be fully monitored under the supervision and care of Dr. Stefany Primeaux in consultation with Dr. Neil Johannsen.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive
2. Fasting glucose above 94 mg/dL and below 125 mg/dl
3. Without diagnosis of diabetes mellitus
4. "No" response to six questions in Physical Activity Readiness Questionnaire (PAR-Q), given at time of screening

Exclusion Criteria:

1. Lack of informed consent
2. Decisionally impaired individuals
3. Non-English speaking
4. Acute illness within the preceding six weeks (defined as fever, new antibiotic use or unscheduled healthcare visit (for illness))
5. Acute alcohol intoxication
6. Pregnancy
7. Currently prescribed blood thinners (if undergoing muscle biopsy)
8. Allergy to Lidocaine (if undergoing muscle biopsy)
9. Significant peripheral neuropathies (if undergoing exercise)
10. Significant cardiovascular impairments (if undergoing exercise)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose and OGTT values (subclinical dysglycemia) | Baseline
  Risk for subclinical dysglycemia

SECONDARY OUTCOMES:
Skeletal muscle phenotype | Baseline
  Subclinical dysglycemia associated with dysfunctional skeletal muscle measured by myomiRs
Fasting plasma glucose | Change from baseline in fasting plasma glucose after 10 weeks
  Glycemic control measured by fasting plasma glucose
myomiRs | Change from baseline in myomiRs after 10 weeks
  Dysfunctional SKM measured by myomiRs

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Molina, MD, PhD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Requests for access to biological samples or existing clinical data obtained from our subjects will be evaluated by Dr. Molina.

REFERENCES:
- [Derived] Primeaux SD, Simon L, Ferguson TF, Levitt DE, Brashear MM, Yeh A, Molina PE. Alcohol use and dysglycemia among people living with human immunodeficiency virus (HIV) in the Alcohol & Metabolic Comorbidities in PLWH: Evidence Driven Interventions (ALIVE-Ex) study. Alcohol Clin Exp Res. 2021 Sep;45(9):1735-1746. doi: 10.1111/acer.14667. Epub 2021 Aug 2. PMID 34342022